CLINICAL TRIAL: NCT04792489
Title: A Multi-center Single Arm Phase II Study to Evaluate the Safety and Efficacy of Genetically Engineered Autologous Cells Expressing Anti-CD20 and Anti-CD19 Specific Chimeric Antigen Receptor in Subjects With Relapsed and/or Refractory Diffuse Large B Cell Lymphoma
Brief Title: DALY II USA/ MB-CART2019.1 for DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2018-344
Record Dates: First submitted 2021-02-25; First posted 2021-03-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Refractory Diffuse Large B Cell Lymphoma (DLBCL); Relapsed Diffuse Large B Cell Lymphoma; High Grade B-cell Lymphoma (HGBCL); Primary Mediastinal B-cell Lymphoma (PMBCL); Transformed Lymphoma; Central Nervous System Lymphoma; Mantle Cell Lymphoma (MCL); Richter Transformation
Keywords: CD19/CD20-directed CAR-T Cells; Zamtocabtagene autoleucel; B-Cell Non-Hodgkin Lymphoma; Primary Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma; NHL; PCNSL; SCNSL; Chimeric Antigen Receptor; CAR; CAR-T Cell; Autologous T Cell Therapy; Central Nervous System Neoplasms; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; MCL; RT; CLL; Immunotherapy; T cells; T cell infusion
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell; Central Nervous System Neoplasms; Lymphoma; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single, open label (Experimental)
  Interventions: Biological: zamtocabtagene autoleucel (MB-CART2019.1); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Bendamustine

INTERVENTIONS:
Biological: zamtocabtagene autoleucel (MB-CART2019.1) — Chimeric antigen receptor (CAR) T cell therapy
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy
Drug: Bendamustine — Lymphodepleting chemotherapy

SUMMARY:
DALY II USA is a phase II, multi-center, single arm study to evaluate the efficacy, safety, and pharmacokinetics of zamtocabtagene autoleucel (MB-CART2019.1) in patients with relapsed and/or refractory diffuse large B cell lymphoma (DLBCL) after receiving at least two lines of therapy. Additional cohorts include subjects with B-cell primary or secondary central nervous system (CNS) lymphoma (PCNSL) and (SCNSL), mantle cell lymphoma (MCL) and Richter's transformation (RT) after receiving at least one line of therapy.

DETAILED DESCRIPTION:
A prospective, single arm, open label, multi-center, phase II study of autologous T cells engineered against both CD19 and CD20 antigens for subjects with relapsed or refractory DLBCL after receiving at least two lines of therapy. The investigational agent is the MB-CART2019.1 cells. Additional cohorts include subjects with B-cell primary or secondary central nervous system (CNS) lymphoma (PCNSL) and (SCNSL), mantle cell lymphoma (MCL) and Richter's transformation (RT) after receiving at least one line of therapy. After successful screening, subjects will undergo leukapheresis to collect product for manufacturing. In preparation for the fresh product infusion, subjects will undergo a lymphodepleting regimen with cyclophosphamide and fludarabine, or bendamustine. Cell infusion will be administered intravenously at a dose of 2.5 x 106 CAR+ cells/kg body weight. The study will start with enrollment of 3 subjects in the lead-in safety phase, and after safety is evaluated, the study will continue with enrollment of the remaining subjects. Subjects will be followed for up to 2 years, for efficacy and safety outcomes as well as health-related quality of life (HRQol). Additional long-term follow-up will be conducted for participants under a separate long-term follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell non-Hodgkin's lymphoma:
* DLBCL DLBCL or associated subtype, defined by WHO 2016 classification:
* DLBCL not otherwise specified (NOS)
* High-grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements
* High-grade B cell lymphoma (NOS)
* Primary mediastinal (thymic) large B cell lymphoma
* Transformed lymphoma (e.g., transformed follicular, or marginal zone lymphoma, follicular lymphoma (FL Grade 3)
* CNS Cohort only: B-cell primary or secondary central nervous system lymphoma (PCNSL or SCNSL)
* Mantle Cell Lymphoma (MCL) Cohort: Histologically confirmed MCL determined by overexpression of cyclin D1 or presence of t(11;14) (q13; q32) translocation
* Richter's Transformation (RT) Cohort: Histologically confirmed Richter's transformation (RT) to a diffuse large B-cell lymphoma (DLBCL) subtype from underlying CLL (clonally related)
* Relapsed or refractory disease is defined for DLBCL (and associated subtypes) population as failure of 2 or more lines of chemotherapy including rituximab or equivalent and anthracycline and either having failed autologous stem cell transplant (ASCT), or ineligible, not intended for or not consenting to ASCT
* Chemotherapy-refractory disease is defined as persistent disease after last line of therapy or relapsed or persistent disease after prior ASCT for lymphoma
* Disease relapse in subjects without prior ASCT is defined as relapse of disease after the last dose of most recent therapy regimen
* CNS Cohort: Subjects with relapsed/refractory PCNSL that have failed (or unable to tolerate) at least first-line therapy.
* No contraindications for MRI evaluation
* CNS Cohort: Subjects with SCNSL must have relapsed or refractory disease after having received at least one prior line of systemic therapy
* Prior lines of systemic therapy should include an anti-CD20 monoclonal antibody and anthracycline containing chemotherapy regimen and/or with or without an autologous stem cell transplant
* No contraindications for MRI evaluation
* MCL Cohort: Subjects with relapsed/refractory disease after at least one prior systemic treatment, that must include:
* Cytotoxic rituximab-based chemotherapy regimen (eg, rituximab bendamustine, R-CHOP, R-DHAP, R-ARA-C) AND
* BTK inhibitor
* RT Cohort: Subject must have relapsed/refractory disease after at least one prior systemic treatment following Richter's Transformation
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening. ECOG performance status of 2 at screen is allowed if the decrease in performance status is due to lymphoma
* Measurable disease according to Lugano 2014 criteria for assessing FDG-PET/CT in systemic lymphoma (Cheson et al, 2014). Measurable disease according to IPCG criteria will be assessed by brain/spine MRI for CNS disease
* Subject must have a tumor biopsy sample (at least 16 unstained slides of tissue or tissue block) from the most recent relapse available prior to MB-CART2019.1 infusion. If medically not feasible to obtain a biopsy from the most recent relapse and for cases when the amount of tissue is limited, the sponsor should be consulted, to confirm adequacy of the sample for study required analyses
* No clinical suspicion of central nervous system (CNS) lymphoma (not applicable to CNS cohort)
* If the subject has history of CNS disease (not applicable to CNS cohort), then he/she must have no signs or symptoms of CNS disease, have no active disease on magnetic resonance imaging (MRI), have no large cell lymphoma present in cerebral spinal fluid (CSF), regardless of the number of white blood cells (WBCs)
* If has history of cerebral vascular accident (CVA), the CVA event must be greater than 12 months prior to leukapheresis. Any neurological deficits must be stable
* A creatinine clearance (as estimated by direct urine collection or Cockcroft-Gault Equation) > 45mL/min
* Cardiac ejection fraction (EF) ≥ 45% as determined by an echocardiogram (ECHO) or Multigated Radionuclide Angiography (MUGA)
* Resting O2 saturation >90% on room air
* Serum alanine aminotransferase (ALT) / aspartate aminotransferase (AST)<5 times the Upper Limit of Normal (ULN) for age
* Total bilirubin <1.5 mg/dl, except in individuals with Gilbert's syndrome
* Absolute neutrophil count (ANC) > 1000/μL
* Absolute lymphocyte count > 100/μL
* Platelet count > 50,000/µL
* Estimated life expectancy of more than 3 months other than primary disease

Exclusion Criteria:

* Primary CNS lymphoma (not applicable to CNS cohort)
* Richter's transformed DLBCL arising from chronic lymphocytic leukemia (CLL) (not applicable to RT cohort)
* Unable to give informed consent
* Known history of infection with human immunodeficiency virus (HIV) or active hepatitis B (HBsAg positive). If there is a history of treated hepatitis B or hepatitis C, the viral load must be quantitative polymerase chain reaction (PCR) negative; antiviral prophylaxis is required if HBsAg negative and anti-HBc positive
* Known history of infection with hepatitis C virus (anti-HCV positive) unless viral load is undetectable per quantitative PCR and/or nucleic acid testing.
* Pharmacologically uncontrolled seizures.
* Known history or presence of autoimmune CNS disease, such as multiple sclerosis, optic neuritis, or other immunologic or inflammatory disease
* Presence of CNS disorder that, in the judgment of the investigator, may impair the ability to evaluate neurotoxicity. For CNS Cohort:
* Midline shift on MRI
* Abnormal high CSF opening pressure and or CSF protein >150 mg/dL Recent (within 3 months) whole brain radiotherapy (WBRT)
* Active systemic fungal, viral, or bacterial infection
* Pregnant or breast-feeding woman
* Previous or concurrent malignancy with the following exceptions:
* Adequately treated basal cell or squamous cell carcinoma (adequate wound healing required prior to study entry)
* In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 2 years prior to the study
* Adequately treated breast or prostate carcinoma on hormonal therapies such as Lupron or tamoxifen and in clinical remission of ≥ 2 years
* A primary malignancy which has been completely resected / treated with curative intent and in complete remission of ≥ 2 years
* Severely immunocompromised subjects e.g., due to current treatment of non-neurologic autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus).
* Medical condition requiring prolonged use of systemic corticosteroids equivalent to prednisone >10 mg/day. For CNS cohort: Up to 2 mg/day dexamethasone (or equivalence) may be allowed at any time, higher doses allowed up to 7 days prior to apheresis or after apheresis until lymphodepletion.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months of enrollment
* Concurrent radiotherapy (normal tissue sparing palliative radiotherapy allowed up to time of lymphodepletion). For systemic therapy, at least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed at the time of scheduled leukapheresis.
* Baseline dementia that would interfere with therapy or monitoring, determined using Immune Effector Cell-Associated Encephalopathy (ICE) Assessment at baseline
* History of severe immediate hypersensitivity reaction to any of the agents used in this study
* Refusal to participate in additional lentiviral gene therapy LTFU protocol
* Prior CAR-T therapy for any indication or systemic gene modifying therapy for B-cell lymphoma
* Prior allogeneic stem cell transplant for any indication
* Prior BITE antibodies for cancer therapy
* Prior T cell receptor-engineered T cell therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | through study completion, up to 2 years
  ORR

SECONDARY OUTCOMES:
Complete Response Rate | 1 and 6 months
  CRR
Duration of Response | Up to 2 years
  DOR
Overall Response Rate | 1 and 6 months
  ORR
Best Overall Response | 2 years
  BOR
Progression Free Survival | Up to 2 years
  PFS
Overall Survival | Up to 2 years
  OS
Type, frequency, and severity of adverse events | Up to 2 years
  Safety
Incidence of anti-MD-CART2019.1 antibodies | Up to 2 years
  Bioanalytical
Phenotype of MB-CART2019.1 | Up to 2 years
  Bioanalytical
Persistence of MB-CART2019.1 | Up to 2 years
  Bioanalytical
Quality of Life (QoL) assessments [EQ-5D-5L] | Up to 2 years
  Health Outcomes - Standardized 5 question measure of health status developed by the EuroQol Group
Patient-Reported Outcome (PRO) assessment [FACT-Lym] | Up to 2 years
  Health Outcomes - To address health-related quality-of-life (HRQL) issues for Non-Hodgkin's lymphoma (NHL) patients
Pharmacodynamics [Levels of cytokines in blood] | Up to 2 years
  Bioanalytical
Correlation of tumor CD19 and CD20 antigen expression with disease progression and relapse | Up to 2 years
  Bioanalytical

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Theruvath, MD, Study Director — Miltenyi Biomedicine GmbH
Locations (25):
- United States (23):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - UC San Diego Health, La Jolla, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - Baptist Health Miami Cancer Institute, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Robert H Lurie Cancer Center, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland Marlene and Stewart Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center - Division of Hematologic Malignancies, Durham, North Carolina
  - The Ohio State University Wexner Medical Center James Cancer, Columbus, Ohio
  - Oregon Health and Science University Knight Cancer Institute, Portland, Oregon
  - Allegheny Health Network Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Alberta Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Miltenyi Biomedicine Website — https://www.miltenyibiomedicine.com/
- See also: Miltenyi Biomedicine DALY II Trial Website — https://www.dalytrials.com/clinical-trial/